CLINICAL TRIAL: NCT03447717
Title: The Long-term Effects of an Implantable Drop Foot Stimulator on Gait in Hemiparetic Patients
Brief Title: Implanted Drop Foot Stimulator for Hemiparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Agnes Sturma, Physitherapist, Researcher, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2126/2016
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Gait, Hemiplegic
Keywords: hemiplegic gait; peroneal nerve stimulation; gait analysis
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: patients meeting the inclusion criteria are included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ActiGait (Experimental): Patients who get the ActiGait implant
  Interventions: Device: ActiGait

INTERVENTIONS:
Device: ActiGait — implanted device for peroneal nerve stimulation

SUMMARY:
The aim of this study is to investigate the effects of the implantable drop foot stimulator "ActiGait" (Ottobock Health Care, Duderstadt, Germany) on gait in hemiparetic patients. While several studies investigated the effects of implanted systems on walking speed and gait endurance, only a few studies have focused on the system's impact on kinematics and long-term outcomes. Therefore, our aim was to further investigate the effects of the implanted system ActiGait on gait kinematics and spatiotemporal parameters with a 1-year follow-up period.

DETAILED DESCRIPTION:
Patients with a neurologic condition leading to drop foot during swing phase in gait are treated by the implentation of the AcitGait system (which has a CE-certificate in Europe).

The aim of this study is to investigate the effect of the device on gait with a follow-up period of one year. Patients are assessed before implantation and at one-year follow up. At baseline, they are asked to walk without any assistive device, as well as with surface electrical stimulation of the peroneal nerve. At follow-up, they are asked to walk with the ActiGait system switched off and switched on.

Outcome assessments include a 10m-walking test and gait analysis with a VICON 3D-camera system. This allows to extract spatio-temporal parameters (as steps per minute, step length,...) as well as kinematic data (e.g. joint ankles during the gait cycle). All outcome data is analyzed using statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* drop foot after stroke, brain haemorrhage or multiple sclerosis
* a minimum of six months after the acute infarction/onset of the disease
* passive extension of the ankle to at least at neutral position
* no sufficient active ankle extension
* free walking without any aid for at least 20 meters in less than 2 minutes
* a walking speed of ≤ 1,2m/sec (measured with 10 meter walking test)
* use of surface electrical stimulation for at least three months
* be able to stand freely

Exclusion Criteria:

* damage to the peripheral nervous system
* epilepsy
* adiposity
* substance abuse
* no cognitive ability to follow the study instructions
* pregnancy
* use of other implanted devices
* instable ankle joint or fixed contracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07-26 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
kinematic gait parameters | 1 year
  Kinematic gait parameters are recorded and analysed using a 3D VICON infra-red camera system.

SECONDARY OUTCOMES:
spatio-temporal parameters | 1 year
  Spatio-temproal parameters are recorded and analysed using a 3D VICON infra-red camera system.
10-m-walking test | 1 year
  The 10-m-walking test is a standardised clinical test where the patient is asked to walk for 10m at the fastest convenient walking speed and time is taken.
Visual Analogue Scale for Health | 1 year
  Using a 100mm Visual Analogue Scale (VAS) patients are asked to mark their current health status between 0 (worst possible health) and 100 (best possible health).

CONTACTS AND LOCATIONS:
Overall Officials: Oskar C Aszmann, MD, Study Director — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: Yes
All IPD from the mentioned outcome parameters are planned to be made available to other researchers.
Time Frame: upon publication in a scientific journal
Access Criteria: publically available